CLINICAL TRIAL: NCT03874403
Title: Advanced Research on the Anesthetic Component and Monitor During the Nonintubated Video-assisted Thoracoscopic Surgery (NIVATS)
Brief Title: Anesthetic Component Research on VATS and NIVATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 201712125RINB
Record Dates: First submitted 2019-02-28; First posted 2019-03-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Thoracoscopy; Anesthesia; Functional; Tracheal Intubation

STUDY DESIGN:
Intervention Model Description: compare the DSA monitoring between the patients receiving intubated or NIVATS
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIVATS (Experimental): Patients receiving Non-intubated VATS with DSA changes
  Interventions: Procedure: DSA
- Intubated VATS (Other): Patients receiving intubated VATS with DSA changes
  Interventions: Procedure: DSA

INTERVENTIONS:
Procedure: DSA — The changes on DSA on NIVATS and VATS

SUMMARY:
The non-intubated video-assisted thoracic surgery (NIVATS) can avoid intubation-related complications and for a smoother postoperative recovery. Successful results are accumulating not only from anecdotal case reports of difficult and high-risk patients not suitable for an intubated general anesthesia. However, in spite of safety and feasibility, there were still three main concerns: 1. how to maintain spontaneous breathing with optimal anesthetic depth; 2. How to analyze the components of general anesthesia and regional anesthesia; 3.what's the benefits on the recovery and the risk of aspiration risk with NIVATS? The traditional monitor or methods such as BIS system, SpO2, and follow-up aspiration signs could not offer sufficient evidence to resolve the three main concerns. Recently, there have been many new methods to monitor these concerns. The density spectral array (DSA) BIS system could analyze the change of the anesthetic component. The ORI is a dimensionless index that reflects oxygenation in the moderate hyperoxic range (PaO2 100-200 mmHg).

DETAILED DESCRIPTION:
Background: The non-intubated video-assisted thoracic surgery (NIVATS) can avoid intubation-related complications and for a smoother postoperative recovery. In recent years, investigator have completed more than 1000 NIVATS. However, the benefits on recovery including swallowing and esophageal function have nerver been demonstrated. The anesthetic components include an intravenous general anesthesia with an intraoperative nerve blocks. Monitoring and analyzing the components of anesthesia have rarely been studied. In this study, the investigator plan to do a radomized control study to demonstarte the differences between NIVATS and intubated VATS, and to investigate the differences on recovery and anesthetic components. Patients schedured for VATS operation, suitable for NIVATS will be included and randomized into NIVATS or VATS groups. DSA and Ce will be monitored throughout the surgical procedures. swalowing test, esophageal function and postoperative qustionare for food intake will be recorded, collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients schedured for VATS operations, suitable for NIVATS after anesthetic evaluation

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The changes of Ce of propofol and remifentanil | four hours in the intraoperative period
  The changes of concentration of effective site (Ce) shown on TCI pump before and after intercostal nerve block in NIVATS and VATS groups
density spectral array changes with thoracoscopic intercostal nerve blocks | four hours in the intraoperative period
  a colour display that represents the frequencies and amplitudes of brain waves through time, with the colour spectrum ranging from blue (minimum amplitude) to dark red (maximum amplitude).

CONTACTS AND LOCATIONS:
Overall Officials: ya-jung Cheng, Study Director — Department of anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan